CLINICAL TRIAL: NCT03466671
Title: An Early Phase II Trial for Efficacy and Safety of TTA-121 on Autism Spectrum Disorder
Brief Title: A Trial of TTA-121 on Autism Spectrum Disorder
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hamamatsu University (Other)
Collaborators: Japan Agency for Medical Research and Development (Other Government)
Responsible Party: Principal Investigator, Hidenori Yamasue, M.D., Ph.D., Professor, Hamamatsu University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMIN000031412
Record Dates: First submitted 2018-02-28; First posted 2018-03-15 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Low dose once per day and placebo (Other): Four weeks administrations of TTA-121 3U once per day in morning and placebo once per day in evening.
  After four weeks washout, four weeks administrations of placebo twice per day in morning and evening.
  Interventions: Drug: TTA-121
- Low dose twice per day and placebo (Other): Four weeks administrations of TTA-121 3U twice per day in morning and evening. After four weeks washout, four weeks administrations of placebo twice per day in morning and evening.
  Interventions: Drug: TTA-121
- High dose once per day and placebo (Other): Four weeks administrations of TTA-121 10U once per day in morning and placebo once per day in evening.
  After four weeks washout, four weeks administrations of placebo twice per day in morning and evening.
  Interventions: Drug: TTA-121
- High dose twice per day and placebo (Other): Four weeks administrations of TTA-121 10U twice per day in morning and evening. After four weeks washout, four weeks administrations of placebo twice per day in morning and evening.
  Interventions: Drug: TTA-121
- Placebo and low dose once per day (Other): Four weeks administrations of placebo twice per day in morning and evening. After four weeks washout, four weeks administrations of TTA-121 3U once per day in morning and placebo once per day in evening.
  Interventions: Drug: TTA-121
- Placebo and low dose twice per day (Other): Four weeks administrations of placebo twice per day in morning and evening. After four weeks washout, four weeks administrations of TTA-121 3U twice per day in morning and evening.
  Interventions: Drug: TTA-121
- Placebo and high dose once per day (Other): Four weeks administrations of placebo twice per day in morning and evening. After four weeks washout, four weeks administrations of TTA-121 10U once per day in morning and placebo once per day in evening.
  Interventions: Drug: TTA-121
- Placebo and high dose twice per day (Other): Four weeks administrations of placebo twice per day in morning and evening. After four weeks washout, four weeks administrations of TTA-121 10U twice per day in morning and evening.
  Interventions: Drug: TTA-121

INTERVENTIONS:
Drug: TTA-121 — A nove intranasal spray of oxytocin and placebo

SUMMARY:
To test efficacy and safety of a novel nasal spray of oxytocin on social deifies in autism spectrum disorder, and To compare effect sizes of different doses

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of autism spectrum disorder based on Diagnostic and Statistical Manual of Mental Disorders-V with score exceeding the cut-off value of 10 for qualitative abnormalities in social reciprocity on Autism Diagnostic Interview Revised (ADIR)
2. Full scale Intelligent quotient above 80 as measured using the Wechsler Adult Intelligent Scale-III
3. Written informed consent for participating the trial

Exclusion Criteria:

1. Diagnosis of bipolar disorder or schizophrenia spectrum disorder
2. Primary diagnosis of depressive disorders, obsessive-compulsive and related disorders, anxiety disorders, trauma- and stressor-related disorders, dissociative disorders, somatic symptom and related disorders, or neurodevelopmental disorders other than autism spectr um disorder
3. Instability in symptoms of comorbid mental disorders such as depressive disorders or anxiety disorders
4. History of changes in medication or doses of psychotropics within one month before registration
5. Current treatment with more than one psychotropics
6. History of hyper-sensitivity to oxytocin
7. History of seizures or traumatic brain injury with loss of consciousness for longer than 5 minutes
8. History of alcohol-related disorders, substance abuse, or addiction
9. Family history of male breast cancer
10. Subject who has severe complications
11. Known hypersensitivity to some drugs and foods
12. Subject who is not able to consent contraception during study period
13. Participation in another registration clinical trial and administration of investigational drug during 120 days before informed consent
14. Other Subjects whom a lead investigator or the patient's primary physician deems are not appropriate for this study

Ages: 18 Years to 54 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2018-02-27 (Actual); Primary Completion 2020-03-16 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy on autism spectrum social core symptom assessed by social reciprocity score on the Autism Diagnostic Observation Schedule module 4 | At baseline, which was before and on the same day as the first administration, and at endpoint, which was started approximately 15 min after the last drug administration
  Changes in social reciprocity score (range: 0-14, Higher value represent a worth outcome) on Autism Diagnostic Observation Schedule module 4 between baseline and endpoint of each administration period

SECONDARY OUTCOMES:
Efficacy on autism spectrum core symptom assessed by communication score on the Autism Diagnostic Observation Schedule module 4 | At baseline, which was before and on the same day as the first administration, and at endpoint, which was started approximately 15 min after the last drug administration
  Changes in communication score (range: 0-8, Higher value represent a worth outcome) on Autism Diagnostic Observation Schedule module 4 between baseline and endpoint of each administration period
Efficacy on autism spectrum core symptom assessed by repetitive and restricted behavior score on the Autism Diagnostic Observation Schedule module 4 | At baseline, which was before and on the same day as the first administration, and at endpoint, which was started approximately 15 min after the last drug administration
  Changes in repetitive and restricted behavior score (range: 0-10, Higher value represent a worth outcome) on Autism Diagnostic Observation Schedule module 4 between baseline and endpoint of each administration period
Efficacy on autism spectrum core symptom assessed by revised algorithm score of social affect on the Autism Diagnostic Observation Schedule module 4 | At baseline, which was before and on the same day as the first administration, and at endpoint, which was started approximately 15 min after the last drug administration
  Changes in revised algorithm score of social affect (range: 0-20, Higher value represent a worth outcome) on Autism Diagnostic Observation Schedule module 4 between baseline and endpoint of each administration period
Efficacy on autism spectrum core symptom assessed by revised algorithm of repetitive and restricted behavior score on the Autism Diagnostic Observation Schedule module 4 | At baseline, which was before and on the same day as the first administration, and at endpoint, which was started approximately 15 min after the last drug administration
  Changes in revised algorithm of repetitive and restricted behavior score (range: 0-10, Higher value represent a worth outcome) on Autism Diagnostic Observation Schedule module 4 between baseline and endpoint of each administration period
Efficacy assessed by Clinical Global Impression-Improvement | At baseline, which was before and on the same day as the first administration, and at endpoint, which was assessed within 100 min after the last drug administration
  Changes in Clinical Global Impression-Improvement (range: 1-7, Higher value represent a worse outcome) between baseline and endpoint of each administration period
Efficacy assessed by Clinical Global Impression-Severity | At baseline, which was before and on the same day as the first administration, and at endpoint, which was assessed within 100 min after the last drug administration
  Changes in Clinical Global Impression-Severity (range: 1-7, Higher value represent a worse outcome) between baseline and endpoint of each administration period
Efficacy assessed by Global Assessment of Functioning | At baseline, which was before and on the same day as the first administration, and at endpoint, which was assessed within 100 min after the last drug administration
  Changes in Global Assessment of Functioning (range: 1-100, Higher value represent a better outcome) between baseline and endpoint of each administration period
Efficacy assessed by gaze fixation time on social region | At baseline, which was before and on the same day as the first administration, and at endpoint, which was started approximately 60 min after the last drug administration
  Changes in gaze fixation time on social region during being talked between baseline and endpoint of each administration period
Efficacy assessed by quantitative analysis of facial expression | At baseline, which was before and on the same day as the first administration, and at endpoint, which was started approximately 15 min after the last drug administration
  Changes in quantitative measure of facial expression on videos recorded during ADOS administration between baseline and endpoint of each administration period

CONTACTS AND LOCATIONS:
Overall Officials: Hidenori Yamasue, MD, PhD, Principal Investigator — Department of Psychiatry, Hamamatsu University School of Medicine
Locations (1):
- Hamamatsu University School of Medicine, Hamamatsu, Shizuoka, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wakuda T, Benner S, Uemura Y, Nishimura T, Kojima M, Kuroda M, Matsumoto K, Kanai C, Inada N, Harada T, Kameno Y, Munesue T, Inoue J, Umemura K, Yamauchi A, Ogawa N, Kushima I, Suyama S, Saito T, Hamada J, Kano Y, Honda N, Kikuchi S, Seto M, Tomita H, Miyoshi N, Matsumoto M, Kawaguchi Y, Kanai K, Ikeda M, Nakamura I, Isomura S, Hirano Y, Onitsuka T, Ozaki N, Kosaka H, Okada T, Kuwabara H, Yamasue H. Oxytocin-induced increases in cytokines and clinical effect on the core social features of autism: Analyses of RCT datasets. Brain Behav Immun. 2024 May;118:398-407. doi: 10.1016/j.bbi.2024.03.013. Epub 2024 Mar 8. PMID 38461957
- [Derived] Yamasue H, Kojima M, Kuwabara H, Kuroda M, Matsumoto K, Kanai C, Inada N, Owada K, Ochi K, Ono N, Benner S, Wakuda T, Kameno Y, Inoue J, Harada T, Tsuchiya K, Umemura K, Yamauchi A, Ogawa N, Kushima I, Ozaki N, Suyama S, Saito T, Uemura Y, Hamada J, Kano Y, Honda N, Kikuchi S, Seto M, Tomita H, Miyoshi N, Matsumoto M, Kawaguchi Y, Kanai K, Ikeda M, Nakamura I, Isomura S, Hirano Y, Onitsuka T, Kosaka H, Okada T. Effect of a novel nasal oxytocin spray with enhanced bioavailability on autism: a randomized trial. Brain. 2022 Apr 18;145(2):490-499. doi: 10.1093/brain/awab291. PMID 35067719